CLINICAL TRIAL: NCT07383623
Title: THE EFFECT OF STAPLER VERSUS SKIN SUTURING ON PAIN AND WOUND HEALING AFTER EPISIOTOMY REPAIR IN PRIMIPAROUS WOMEN: A RANDOMIZED CONTROLLED TRIAL
Brief Title: THE EFFECT OF STAPLER VERSUS SKIN SUTURING ON PAIN AND WOUND HEALING AFTER EPISIOTOMY REPAIR IN PRIMIPAROUS WOMEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşegül Kanık (Other)
Responsible Party: Sponsor-Investigator, Ayşegül Kanık, MIDWIFE, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THESIS-EPIS-PAIN-2025
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Episiotomy
Keywords: episiotomy; stapler; primiparous women

STUDY DESIGN:
Intervention Model Description: Primiparous women are randomly assigned to one of two parallel groups to undergo episiotomy repair with either stapler or absorbable skin sutures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stapler skin closure group (Experimental): Episiotomy repair is performed using surgical staplers for skin closure in primiparous women.
  Interventions: Device: stapler skin closure
- Absorbable suture group (Experimental): Skin closure of episiotomy is performed using absorbable sutures.
  Interventions: Procedure: absorbable suture group

INTERVENTIONS:
Device: stapler skin closure — skin closure of episiotomy is performed using a surgical stapler.
  Arms: stapler skin closure group
Procedure: absorbable suture group — skin closure of episiotomy is performed using absorbable sutures.
  Arms: Absorbable suture group

SUMMARY:
This randomized controlled study aims to evaluate the effects of skin closure using surgical staplers compared with conventional skin sutures on postoperative pain and wound healing in primiparous women undergoing episiotomy repair after vaginal delivery.

Primiparous women who require episiotomy during vaginal birth will be randomly assigned to one of two groups: skin closure with staples or skin closure with sutures. Postpartum pain levels and wound healing outcomes will be assessed and compared between the two groups.

The results of this study are expected to contribute to evidence-based decisions regarding optimal skin closure techniques in episiotomy repair.

DETAILED DESCRIPTION:
Episiotomy is one of the most commonly performed obstetric interventions during childbirth. Although it shares similar characteristics with spontaneous second-degree perineal tears, episiotomy was routinely performed for many years. However, routine episiotomy practices began to be questioned in the late 1970s and 1980s, and its use declined during the 1990s. Factors contributing to this change include increased health awareness among women, the natural childbirth movement, professional competition, and the widespread adoption of evidence-based practices.

Pain associated with episiotomy is a significant issue that negatively affects women's quality of life in the postpartum period. A woman's request for analgesia is considered a medical indication for pain management. Inadequate pain control reduces the effectiveness of therapeutic interventions. Episiotomy-related pain decreases maternal comfort, negatively affects mother-infant bonding, reduces breastfeeding success, and may even influence women's childbirth preferences due to fear of labor and episiotomy pain.

The ideal method for episiotomy repair should be fast, easy to perform, cause minimal tissue trauma, and result in minimal postpartum pain and dyspareunia. Closure techniques that minimize skin trauma reduce inflammation and scarring by limiting the introduction of foreign materials. Various techniques have been proposed for postpartum episiotomy repair, including non-suturing of the incision, continuous locking sutures, and interrupted non-locking sutures. Regardless of the technique used, successful tissue approximation is associated with less pain and wound infection, better cosmetic outcomes, and shorter hospital stays.

In recent years, traditional repair methods have increasingly been replaced by modern techniques such as skin staples, tissue adhesives, and adhesive strips. Skin staples, one of these modern methods, are described as a faster and more reliable repair technique. Due to their fixed depth and uniform structure, staples provide equal wound tension, which is thought to reduce pain and promote wound healing in episiotomy skin repair.

The aim of this study is to determine the effects of using staples versus surgical sutures in episiotomy skin repair on postpartum localized pain and wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Term pregnancy (≥ 37 weeks)
* Low-risk pregnancy (no obstetric risk factors)
* Not receiving oxytocin induction during latent or active labor
* Singleton pregnancy with a live fetus
* No psychiatric disorder
* No substance abuse
* Primiparous women (first vaginal birth)
* Presence of 1st or 2nd degree perineal tear
* Able to read, understand, and voluntarily provide written and verbal informed consent.

Exclusion Criteria:

* Apgar score < 7 at 1 minute and/or 5 minutes
* Neonatal anomaly
* Use of >10 mL analgesic during episiotomy repair beyond routine practice
* Obesity
* Vaginal infection or vaginal lesion
* Maternal conditions impairing wound healing (e.g., diabetes mellitus, immunosuppression, coagulation disorders)
* 3rd or 4th degree perineal tear
* Shoulder dystocia / difficult delivery

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study includes primiparous women who have undergone vaginal delivery with mediolateral episiotomy.
Enrollment: 24 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
postpartum perineal pain | At 6 hours, 24 hours and 7 days postpartum
  Perineal pain severity will be assessed using the Visual Analog Scale (VAS) following episiotomy repair. The VAS ranges from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Higher scores indicate worse pain severity.

SECONDARY OUTCOMES:
Episiotomy wound healing | 10 days postpartum
  Wound healing will be assessed using the REEDA scale (Redness, Edema, Ecchymosis, Discharge, Approximation). The total REEDA score ranges from 0 to 15, with lower scores indicating better wound healing and higher scores indicating worse wound healing.Wound healing assessed using the REEDA scale (Redness, Edema, Ecchymosis, Discharge, Approximation)

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Demokrasi Universitesi Buca Seyfi Demirsoy Egitim ve Arastirma Hastanesi, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to patient confidentiality and ethical considerations.

REFERENCES:
- [Background] Teixeira, T. T., Caroci-Becker, A., Brunelli, W. S., & Riesco, M. L. G. (2020). Tissue Adhesive To Repair First-Degree Perineal Tear: A Pilot Randomized Controlled Trial. Clinical And Experimental Obstetrics And Gynecology, 47(2), 228-233.
- [Background] Swenson, C. W., Low, L. K., Kowalk, K. M., & Fenner, D. E. (2019). Randomized Trial Of 3 Techniques Of Perineal Skin Closure During Second-Degree Perineal Laceration Repair. Journal Of Midwifery & Women's Health, 64(5), 567-577.
- [Background] Woldegeorgis, B. Z., Obsa, M. S., Tolu, L. B., Bogino, E. A., Boda, T. I., & Alemu, H. B. (2022). Episiotomy Practice and Its Associated Factors in Africa: A Systematic Review and Meta-Analysis. Frontiers in Medicine, 1714.
- [Background] Sherif, A., & El-Shourbagy, M. (2020). Skin-Adhesive Tape Versus Interrupted Suture İn Episiotomy Skin Repair: Randomized Control Trial. Open Journal Of Obstetrics And Gynecology, 10(02), 254.
- [Background] Shahrahmani, H., Kariman, N., Jannesari, S., Rafieian-Kopaei, M., Mirzaei, M., Ghalandari, S., ... & Mardani, G. (2018). The Effect Of Green Tea Ointment On Episiotomy Pain And Wound Healing in Primiparous Women: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Phytotherapy Research, 32(3), 522-530.
- [Background] JahaniShoorab, N., Zagami, S. E., Nahvi, A., Mazluom, S. R., Golmakani, N., Talebi, M., & Pabarja, F. (2015). The effect of virtual reality on pain in primiparity women during episiotomy repair: a randomize clinical trial. Iranian journal of medical sciences, 40(3), 219.
- [Background] Mastud, K., Lamture, Y., Nagtode, T., & Rewale, V. (2022). A Comparative Study Between Conventional Sutures, Staples, And Adhesive Glue For Clean Elective Surgical Skin Closure. Cureus, 14(11).
- [Background] Figueroa, D., Jauk, V. C., Szychowski, J. M., Garner, R., Biggio, J. R., Andrews, W. W., ... & Tita, A. T. (2013). Surgical Staples Compared With Subcuticular Suture For Skin Closure After Cesarean Delivery: A Randomized Controlled Trial. Obstetrics And Gynecology, 121(1).
- [Background] Feigenberg, T., Maor-Sagie, E., Zivi, E., Abu-Dia, M., Ben-Meir, A., Sela, H. Y., & Ezra, Y. (2014). Using Adhesive Glue To Repair First Degree Perineal Tears: A Prospective Randomized Controlled Trial. Biomed Research International, 2014.
- [Background] Corrêa, M. D., & Passini, R. (2016). Selective episiotomy: indications, techinique, and association with severe perineal lacerations. Revista Brasileira de Ginecologia e Obstetrícia, 38(06), 301-307.
- [Background] Deyaso, Z. F., Chekole, T. T., Bedada, R. G., Molla, W., Uddo, E. B., & Mamo, T. T. (2022). Prevalence of Episiotomy Practice and Factors Associated with it in Ethiopia, Systematic Review and Meta-analysis. Women's Health, 18, 17455057221091659.
- [Background] Chang, S. R., Chen, K. H., Lin, H. H., Chao, Y. M. Y., & Lai, Y. H. (2011). Comparison Of The Effects Of Episiotomy And No Episiotomy On Pain, Urinary İncontinence, And Sexual Function 3 Months Postpartum: A Prospective Follow-Up Study. International Journal Of Nursing Studies, 48(4), 409-418.
- [Background] Chamariya, S., Prasad, M., & Chauhan, A. (2016). Comparison Of Dermabond Adhesive Glue With Skin Suture For Repair Of Episiotomy. International Journal Of Reproduction, Contraception, Obstetrics And Gynecology, 5(10), 3461-3466.
- [Background] Akopov, A., Artioukh, D. Y., & Molnar, T. F. (2021). Surgical Staplers: The History Of Conception And Adoption. The Annals Of Thoracic Surgery, 112(5), 1716-1721.
- [Background] Beşen, M. A., & Rathfısch, G. (2019). Doğumda Perineal Travma ve Onarımı: Kanıt Temelli Yaklaşımlar. Gazi Sağlık Bilimleri Dergisi, 4(3), 1-11.